CLINICAL TRIAL: NCT03554187
Title: Efficacy of Supplementation With Probiotics as Adjuvant to Mechanical Treatment in Chronic Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PiLeJe (Industry)
Responsible Party: Sponsor
Organization: Larena SAS (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pil-Clin-BuccP-016; 2017-A02945-48 (Other: Number ID-RCB)
Record Dates: First submitted 2018-03-16; First posted 2018-06-13 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2020-09

CONDITIONS: Probiotics, Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactibiane Buccodental, probiotics (Experimental): For one tablet : Lactobacillus paracasei LA 802 (109 UFC), Vitamine D3 (1,5 µg), Vitamine C (24 mg) Dosage : 2 tablets daily for 6 weeks tablet to suck after the meal and brushing teeth (one in the morning and one in the evening)
  Interventions :
  Ultrasonic periodontal debridement, with appropriate device : D+1 / Analyzes of periodontopathogenic bacteria : D-14, D+1, D+45, D+90 / IL1B test : D-14 / Salivary sampling : D+1, D+45, D+90 / Halitosis measure : D+1, D+45, D+90
  Interventions: Device: Ultrasonic periodontal Debridement, with appropriate device; Biological: Analyzes of periodontopathogenic bacteria; Genetic: IL1B test; Biological: Salivary Sampling; Device: Halitosis measure
- Placebo (Placebo Comparator): With no metabolic action ; identical in appearance to experimental probiotics Dosage : 2 placebo tablets daily for 6 weeks tablet to suck after the meal and brushing teeth (one in the morning and one in the evening)
  Intervention(s) :
  Ultrasonic periodontal debridement, with appropriate device : D+1 / Analyzes of periodontopathogenic bacteria : D-14, D+1, D+45, D+90 / IL1B test : D-14 / Salivary sampling : D+1, D+45, D+90 / Halitosis measure : D+1, D+45, D+90
  Interventions: Device: Ultrasonic periodontal Debridement, with appropriate device; Biological: Analyzes of periodontopathogenic bacteria; Genetic: IL1B test; Biological: Salivary Sampling; Device: Halitosis measure

INTERVENTIONS:
Device: Ultrasonic periodontal Debridement, with appropriate device — Dental procedure that includes therapeutic interventions such as scaling to remove calculus and all soft deposits, root planing to eliminate subgingival calculus and smooth the tooth surface, and root débridement to eliminate subgingival biofilm and lightly mineralized deposits.
Biological: Analyzes of periodontopathogenic bacteria — Collection of plaque, to analyze the bacteria in the pocket
Genetic: IL1B test — susceptibility to periodontal disease (scratch swab onto the tongue) (no invasive)
Biological: Salivary Sampling — Salivette to chew. To analyse salivary microbiota
Device: Halitosis measure — With appropriate device : halimeter

SUMMARY:
It aims to demonstrate the superiority of a 6-week supplementation with Lactibiane Buccodental compared to placebo, as adjunctive therapy in chronic periodontitis in patients with generalized chronic periodontitis

ELIGIBILITY:
Inclusion criterion:

* Age ≥ 18;
* Patient with moderate to severe chronic periodontitis (mean attachment loss ≥ 3 mm), generalized (more than 30% of sites with loss of attachment), with presence of at least one of three bacterial species the red complex (either Pg, Tf or Td), which, according to the practitioner, may be the result of mechanical treatment (ultrasonic debridement);
* Patient able and willing to participate in the research by complying with the procedures of the protocol especially concerning the consumption of the product under study and having served it by signing a dated informed consent form;

Criteria of non-inclusion:

* Patient with acute oral lesions or necrotizing ulcerative periodontitis;
* Patient who has taken antibiotics in the last 3 months, or who has received treatment affecting periodontal tissue in the past month, or on immunosuppressive therapy (ciclosporin), antihypertensive (nyfedipine), antiepileptic (phenytoin), under biotherapy, or under treatment of hyposialie;
* Patient with a medical history or current pathology that, in the opinion of the investigator, is likely to interfere with the results of the study or to expose him / her to additional risk: unbalanced diabetes, rheumatic fever, disease affecting renal or hepatic function, neurological deficiency, immunological disease;
* Patient smoking more than 10 cigarettes a day;
* Patient with known allergy to at least one of Lactibiane Buccodental® ingredients;
* Pregnant or breastfeeding woman or intending to start a pregnancy within 3 months;
* a woman who is in a state of childbearing not covered by an active method of contraception;
* Patient with a psychological or linguistic disability to understand and sign informed consent, or to understand and implement the constraints of the study;
* Patient participating in another clinical trial, or at the time of exclusion from another clinical trial;
* Patient under legal protection (tutorship, guardianship) or deprived of his rights following the administrative or judicial decision.
* Patient not affiliated to a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
Mean level of clinical attachment (CAL) | up to 3 months
  Clinical Attachment (CAL) of parondontal pocket ; measurement with Florida Probe in millimeters

SECONDARY OUTCOMES:
Quantitative evolution of Aggregatibacter actinomycetemcomitans (Aa) bacteria | day -14, day 1, day 45, day 90
  measured from a non-invasive sample in the parontal pocket. Result expressed in number of bacteria
Quantitative evolution of Porphyromonas gingivalis (Pg) bacteria | day -14, day 1, day 45, day 90
  measured from a non-invasive sample in the parontal pocket. Result expressed in number of bacteria
Quantitative evolution of Tannerella forsythia (Tf) bacteria | day -14, day 1, day 45, day 90
  measured from a non-invasive sample in the parontal pocket. Result expressed in number of bacteria
Quantitative evolution of Treponema denticola (Td) bacteria | day -14, day 1, day 45, day 90
  measured from a non-invasive sample in the parontal pocket. Result expressed in number of bacteria
Quantitative evolution of Prevotella intermedia (Pi) bacteria | day -14, day 1, day 45, day 90
  measured from a non-invasive sample in the parontal pocket. Result expressed in number of bacteria
Quantitative evolution of Fusobacterium nucleatum (Fn) bacteria | day -14, day 1, day 45, day 90
  measured from a non-invasive sample in the parontal pocket. Result expressed in number of bacteria
Evolution of several oral indices : Pocket depth | day -14, day 1, day 45, day 90
  pocket depth in millimeters (measured with Florida Probe)
Evolution of several oral indices : Gingival recession | day -14, day 1, day 45, day 90
  gingival recession in millimeters (measured with Florida Probe)
Evolution of several oral indices : Gingival bleeding on probing | day -14, day 1, day 45, day 90
  gingival bleeding on probing (Florida Probe) in percentage
Evolution of halitosis | day -14, day 1, day 45, day 90
  In expired breath : Volatil Sulfur Compounds (in ppm) measure with Halimeter
Overall clinical course of periodontitis | day -14, day 1, day 45, day 90
  according to the dentist, in habitual practise
Safety (tolerance to treatment) | up to a year
  calculated with adverse events that may be observed during study period (descriptif results)
Evaluate adherence to treatment | up to a year
  Quick estimation at D+90

CONTACTS AND LOCATIONS:
Overall Officials: Samira Ait Abdellah, Study Director — PiLeJe
Locations (2):
- France (2):
  - CHU Service d'Odontologie, Lyon, Auvergne-Rhône-Alpes
  - CHU Hôtel Dieu de Nantes, Nantes, Pays de la Loire Region

IPD SHARING:
Plan to Share IPD: No